CLINICAL TRIAL: NCT03128749
Title: Mindfulness-Based Cognitive Therapy: Efficacy and fMRI-based Response Predictors in a Group of OCD Patients Non-responders to CBT
Brief Title: Mindfulness-Based Cognitive Therapy: Efficacy and fMRI-based Response Predictors in a Group of OCD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Hospital Universitari de Bellvitge (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Arizona (Other)
Responsible Party: Principal Investigator, Clara López-Solà, PhD, Corporacion Parc Tauli
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CorporacionPT CIR2016/030
Record Dates: First submitted 2017-04-07; First posted 2017-04-25 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Mindfulness Based Intervention; Cognitive-Behavioral Therapy; Functional Magnetic Resonance Imaging; Neuropsychology; Childhood Maltreatment
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Intervention (Experimental): Mindfulness-based cognitive therapy (MBCT), adjusted to OCD patients, will be applied in 10 weekly sessions of 2 hours followed by an extra session 4 weeks later. The treatment will be applied in a group format of 10 to 12 patients.
  These patients will be also attending to their regular psychiatric visits for medication control.
  Interventions: Behavioral: Mindfulness Based Intervention; Drug: Treatment as Usual
- Treatment as Usual (TAU) (Active Comparator): Patients will be attending to their regular psychiatric visits during the whole trial period.
  Interventions: Drug: Treatment as Usual

INTERVENTIONS:
Behavioral: Mindfulness Based Intervention — The mindfulness based intervention protocol used in this project is adapted from the original and validated MBCT program for depression (Segal, Williams & Teasdale, 2002). Two more sessions, focused on obsessive symptoms specfic to each participant, will be included. Those two sessions will be adapted from the manual "The Mindfulness Workbook for OCD" (Hershfield and Corboy, 2013).
  Other Names: MBCT
  Arms: Mindfulness Based Intervention
Drug: Treatment as Usual — The psychiatric referee will follow OCD guidelines modifying or potentiating drug treatments if needed.
  Other Names: TAU

SUMMARY:
Obsessive-Compulsive Disorder (OCD) patients have a response rate of 50-60% to exposure and response prevention (ERP) therapy and SSRI antidepressants. Mindfulness-Based Cognitive Therapy (MBCT) consists of training the participant to non-react to negative thoughts and emotions. Applying MBCT to OCD patients may help them behave with equanimity in response to their obsessions, and therefore acknowledge them with the same attention and intention as they admit any other disturbing thought without reacting to it. MBCT has demonstrated effectiveness in major depression, but much less attention has been given to MBCT in OCD. ERP and MBCT, although sharing aspects like exposure, are based on different theoretic and therapeutic factors. EPR is based on a direct anxiety habituation process whereas MBCT trains a holistic manner of becoming familiarized with distressful thoughts and emotions while learning to develop a new relationship to them. Thus, MBCT may decrease anxiety indirectly through a major attention awareness and non-reactivity to thoughts and emotions.

OCD is characterized by altered cortical-striatal-thalamic-cortical (CSTC) circuit and default mode network (DMN) connectivity when performing different tasks and during the resting state. It has been establish that the ventral CSTC circuit is mostly associated with emotional processing, while the dorsolateral aspect of the CSTC circuit is preferentially involved in cognitive processing. In this regard, we hypothesized that clinical amelioration will be accompanied by a re-establishment of functional connectivity within dorsolateral and DMN circuits, which will in turn be associated with improvement of certain neuropsychological processes. CSTC and DMN circuits have also shown to be sensitive to prolonged stress situations. Specifically, childhood trauma has been related to larger brain volumes and it has been associated with different OCD clinical subtypes.

Aims: 1. To assess MBCT effectiveness in treatment non-naive OCD patients. 2. To study cognitive and neuropsychological characteristics that mediate or moderate MBCT response. 3. To examine the changes in cognitive, neuropsychological and neuroimaging patterns associated with an MBCT intervention. 4. To identify a brain biomarker for positive response to MBCT in non-naïve OCD patients. 5. To study cognitive, neuropsychological and early stress expousure mediators or moderators of functional changes in CSTC and DMN patterns in response to MBCT.

ELIGIBILITY:
Inclusion Criteria:

* Age frame: 18-50 years old.
* Principal Diagnosis: Obsessive compulsive disorder.
* Severity of OCD symptoms: between mild (Y-BOCS=9) and severe (Y-BOCS=32)
* Previous structured CBT or EPR, either in group or individual format, between 10 to 20 sessions.
* A maximum of three different pharmacological strategies.
* Minimum of IQ 85 measured by Vocabulary subtest (WAIS-IV).
* Minimum level of schooling: 14 years.
* To sign the informant consent.

Exclusion Criteria:

* Organic pathology and/or neurological disorders such as brain injury or epilepsy.
* Comorbidity with: Mental Retardation, previous or current substance abuse, psychotic disorders, bipolar disorder. Other affective and/or anxiety disorders will not be an exclusion criteria if OCD is considered the primary diagnosis.
* Recent suicide attempt/active suicidality
* Previous completion of an MBCT course (≥ 8 weeks)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Y-BOCS: | Baseline and at 14 weeks and at 6 months post-treatment
  • Clinical version of the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) the severity and the checklist.
Change in OCI-R: | Baseline, at 14 weeks and at 6 months post-treatment
  • Obsessive-Compulsive Inventory-Revised (OCI-R) assessing 6 dimensions (Washing, Checking, Ordering, Obsessing, Hoarding and Neutralizing).
Change in OBQ-44: | Baseline and at 14 weeks
  • Obsessive Beliefs Questionnaire-44 (OBQ-44), a measure of three OCD-related belief domains (Perfectionism/Certainty, Importance/Control of thoughts, and Responsibility/Threat estimation).
Changes in functional brain circuits: | Baseline and at 14 weeks
  • Functional Magnetic Resonance Imaging: Resting state and during task performance (Autobiographical memory + N-Back) and self-reference.

SECONDARY OUTCOMES:
Change in anxiety: | Baseline and at 14 weeks
  • Anxiety Sensitivity Index (ASI-3)
Change in mood from baseline: | Baseline, at 14 weeks and at 6 months post-treatment
  • The Beck Depression Inventory (BDI-II)
Change in positive and negative affect: | Baseline and at 14 weeks
  • Positive and Negative Affect trait (PANAS)
Impact of current life events: | Baseline, 14 weeks and at 6 months post-treatment
  • Perceived Stress Scale (PSS)
Impact of past stressful life events: | Baseline
  • Childhood Trauma Questionnaire (CTQ)
Change in attentional domains: | Baseline and at 14 weeks
  • Conners' Continuous Performance Test II : CPT-II
Change in executive Functioning/Cognitive flexibility: | Baseline and at 14 weeks
  • Wisconsin Card Sorting Test: WCST
Autobiographical memories: | Baseline
  • Autobiographic Memory Task: 10 selected emotions (5 negative and 5 positive).
Change in verbal fluency: | Baseline, 14 weeks and at 6 months post-treatment
  • Phonetic Fluency: PMR (Spanish version of the FAS)
Speech analysis: | Baseline
  • Word Task: Assessment of language fluency and thought content using a list of 10 seed words from the Spanish adaptation of the ANEW (Affective Norms for English Words) in terms of positive and negative valance and different degrees of arousal.
Thought content: | Baseline, each week during the treatment period (10 sessions) and post-treatment
  • ES-Questionnaire, designed by Drs. J. Andrews-Hanna and M. López-Solà (research collaborators of the project) from the USA. It is based on 23 questions that examines the thought content from the patient before, during and after the treatment.
Change in Quality of Life: | Baseline, 14 weeks and at 6 months post-treatment
  • Multicultural Quality of Life Index (MQLI).
Change in Mindfulness variables: | Baseline, 14 weeks and at 6 months post-treatment
  • Mindfulness measures include: The Five Facet Mindfulness Questionnaire (FFMQ), used to measure the five constructs central to mindfulness (Observing, Describing, Acting with Awareness, Non-judgment of Inner Experience, and Non-reactivity to Inner Experience).
Change in Rumination: | Baseline, 14 weeks and at 6 months post-treatment
  • Ruminative Responses Scale (RRS) to measure the degree and type of thought thinking.
Treatment expectancy: | Baseline
  • Credibility Expectancy Questionnaire (CEQ).
Changes in structural brain regions: | Baseline and at 14 weeks
  • Structural acquisition: T13D

CONTACTS AND LOCATIONS:
Overall Officials: Clara López-Solà, PhD, Principal Investigator — Corporació Parc Taulí; Maria Serra-Blasco, PhD, Principal Investigator — Fundació Parc Taulí; Pino Alonso, MD, PhD, Principal Investigator — Bellvitge University Hospital; Marina López-Solà, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Jessica Andrews-Hanna, PhD, Principal Investigator — University of Arizona
Locations (1):
- Corporacion Sanitaria Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weissman MM, Bland RC, Canino GJ, Greenwald S, Hwu HG, Lee CK, Newman SC, Oakley-Browne MA, Rubio-Stipec M, Wickramaratne PJ, et al. The cross national epidemiology of obsessive compulsive disorder. The Cross National Collaborative Group. J Clin Psychiatry. 1994 Mar;55 Suppl:5-10. PMID 8077177
- [Background] Murray CJ, Lopez AD. Evidence-based health policy--lessons from the Global Burden of Disease Study. Science. 1996 Nov 1;274(5288):740-3. doi: 10.1126/science.274.5288.740. No abstract available. PMID 8966556
- [Background] Lopez-Sola C, Fontenelle LF, Verhulst B, Neale MC, Menchon JM, Alonso P, Harrison BJ. DISTINCT ETIOLOGICAL INFLUENCES ON OBSESSIVE-COMPULSIVE SYMPTOM DIMENSIONS: A MULTIVARIATE TWIN STUDY. Depress Anxiety. 2016 Mar;33(3):179-91. doi: 10.1002/da.22455. Epub 2015 Dec 2. PMID 26630089
- [Background] Rufer M, Fricke S, Moritz S, Kloss M, Hand I. Symptom dimensions in obsessive-compulsive disorder: prediction of cognitive-behavior therapy outcome. Acta Psychiatr Scand. 2006 May;113(5):440-6. doi: 10.1111/j.1600-0447.2005.00682.x. PMID 16603035
- [Background] Mataix-Cols D, Marks IM, Greist JH, Kobak KA, Baer L. Obsessive-compulsive symptom dimensions as predictors of compliance with and response to behaviour therapy: results from a controlled trial. Psychother Psychosom. 2002 Sep-Oct;71(5):255-62. doi: 10.1159/000064812. PMID 12207105
- [Background] Whittal ML, Robichaud M, Thordarson DS, McLean PD. Group and individual treatment of obsessive-compulsive disorder using cognitive therapy and exposure plus response prevention: a 2-year follow-up of two randomized trials. J Consult Clin Psychol. 2008 Dec;76(6):1003-14. doi: 10.1037/a0013076. PMID 19045968
- [Background] Houghton S, Saxon D, Bradburn M, Ricketts T, Hardy G. The effectiveness of routinely delivered cognitive behavioural therapy for obsessive-compulsive disorder: a benchmarking study. Br J Clin Psychol. 2010 Nov;49(Pt 4):473-89. doi: 10.1348/014466509X475414. Epub 2009 Oct 21. PMID 19849894
- [Background] Jain S, Shapiro SL, Swanick S, Roesch SC, Mills PJ, Bell I, Schwartz GE. A randomized controlled trial of mindfulness meditation versus relaxation training: effects on distress, positive states of mind, rumination, and distraction. Ann Behav Med. 2007 Feb;33(1):11-21. doi: 10.1207/s15324796abm3301_2. PMID 17291166
- [Background] Benzina N, Mallet L, Burguiere E, N'Diaye K, Pelissolo A. Cognitive Dysfunction in Obsessive-Compulsive Disorder. Curr Psychiatry Rep. 2016 Sep;18(9):80. doi: 10.1007/s11920-016-0720-3. PMID 27423459
- [Background] Chiesa A, Anselmi R, Serretti A. Psychological mechanisms of mindfulness-based interventions: what do we know? Holist Nurs Pract. 2014 Mar-Apr;28(2):124-48. doi: 10.1097/HNP.0000000000000017. PMID 24503749
- [Background] Radua J, Mataix-Cols D. Voxel-wise meta-analysis of grey matter changes in obsessive-compulsive disorder. Br J Psychiatry. 2009 Nov;195(5):393-402. doi: 10.1192/bjp.bp.108.055046. PMID 19880927
- [Background] Menzies L, Chamberlain SR, Laird AR, Thelen SM, Sahakian BJ, Bullmore ET. Integrating evidence from neuroimaging and neuropsychological studies of obsessive-compulsive disorder: the orbitofronto-striatal model revisited. Neurosci Biobehav Rev. 2008;32(3):525-49. doi: 10.1016/j.neubiorev.2007.09.005. Epub 2007 Oct 17. PMID 18061263
- [Background] Beucke JC, Sepulcre J, Eldaief MC, Sebold M, Kathmann N, Kaufmann C. Default mode network subsystem alterations in obsessive-compulsive disorder. Br J Psychiatry. 2014 Nov;205(5):376-82. doi: 10.1192/bjp.bp.113.137380. Epub 2014 Sep 25. PMID 25257066
- [Background] Gottlich M, Kramer UM, Kordon A, Hohagen F, Zurowski B. Resting-state connectivity of the amygdala predicts response to cognitive behavioral therapy in obsessive compulsive disorder. Biol Psychol. 2015 Oct;111:100-9. doi: 10.1016/j.biopsycho.2015.09.004. Epub 2015 Sep 18. PMID 26388257
- [Background] Segal ZV, Williams JMG, Teasdale JD (2002) Mindfulness-based cognitive therapy for depression: a new approach to preventing relapse. Guilford, New York.
- [Background] Brooks SJ, Naidoo V, Roos A, Fouche JP, Lochner C, Stein DJ. Early-life adversity and orbitofrontal and cerebellar volumes in adults with obsessive-compulsive disorder: voxel-based morphometry study. Br J Psychiatry. 2016 Jan;208(1):34-41. doi: 10.1192/bjp.bp.114.162610. Epub 2015 Sep 3. PMID 26338992
- [Background] Lochner C, du Toit PL, Zungu-Dirwayi N, Marais A, van Kradenburg J, Seedat S, Niehaus DJ, Stein DJ. Childhood trauma in obsessive-compulsive disorder, trichotillomania, and controls. Depress Anxiety. 2002;15(2):66-8. doi: 10.1002/da.10028. PMID 11891995
- [Background] Goldberg X, Soriano-Mas C, Alonso P, Segalas C, Real E, Lopez-Sola C, Subira M, Via E, Jimenez-Murcia S, Menchon JM, Cardoner N. Predictive value of familiality, stressful life events and gender on the course of obsessive-compulsive disorder. J Affect Disord. 2015 Oct 1;185:129-34. doi: 10.1016/j.jad.2015.06.047. Epub 2015 Jul 2. PMID 26172984
- [Derived] Miquel-Giner N, Vicent-Gil M, Martinez-Zalacain I, Porta-Casteras D, Mar L, Lopez-Sola M, Andrews-Hanna JR, Soriano-Mas C, Menchon JM, Cardoner N, Alonso P, Serra-Blasco M, Lopez-Sola C. Efficacy and fMRI-based response predictors to mindfulness-based cognitive therapy in obsessive-compulsive disorder: Study protocol for a randomised clinical trial. Span J Psychiatry Ment Health. 2023 January/March;18(1):6-12. doi: 10.1016/j.rpsm.2022.11.002. Epub 2022 Nov 17. English, Spanish. PMID 37839958